CLINICAL TRIAL: NCT00243451
Title: Early Detection of Mild Cognitive Impairment in Individual Patients
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, James C. Patterson, II, MD. Ph, Professor, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: LSUHSC H04-049
Record Dates: First submitted 2005-09-13; First posted 2005-10-24 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Mild Cognitive Impairment; Mild Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PET scan & fMRI — Subjects will be screened and if applicable for the study will be scheduled for an MRI. At the third visit they will complete the PET scan. They will return at 6, 12, 24, and 36 months and complete another PET scan at the last visit.

SUMMARY:
Our central hypothesis is that the early metabolic lesions of MCI can be reliably detected in individual subjects by objective analysis of [18]F-fluorodeoxyglucose (FDG) positron-emission tomography (PET) brain images, earlier and more accurately than by subjective clinician rating.

DETAILED DESCRIPTION:
Our goal with this proposal is a prospective, longitudinal study that will examine subjects over a three-year span to establish the presence of MCI, evaluate progression of disease, and determine the validity of this method in detecting early MCI. Specifically, we predict that by using our Cognitive Decline Index (CDI) method of objective examination of FDG PET brain images from patients diagnosed with MCI or mild AD, we can accurately discriminate very early abnormalities in cerebral metabolism, and that this research method can be validated and translated into a clinically useful tool for the early detection of MCI. Our long-range goals are the development of methods and tools that enable the detection of pathology in individual patients at risk for cognitive impairment.

ELIGIBILITY:
MCI Inclusion Criteria (patients):

MCI criteria met:

1. Memory complaint, preferably corroborated by an informant.
2. Objective memory impairment (based on cognitive test scores).
3. Normal general cognitive function.
4. Intact ADL.
5. Not demented.

   * At least 10 years of education, or GED, or equivalent.
   * Patients with ApoE4 positive homozygous or heterozygous status and/or first-degree relative with probable AD are preferred, but patients who meet all other criteria including well-defined MCI criteria will be accepted.
   * Age: 55-85
   * Have normal or clinically unimportant physical exam, beyond those consistent with a diagnosis of MCI.
   * Able to give informed consent, or assent and informed consent from a legal representative.
   * Centrally acting medications will be closely tracked, patients on any such medications will be PET-scanned only after a 24-hour washout, with meds restarted immediately after the scan.
   * Because depression and depressive pseudodementia are often prodromal to cognitive decline, these diagnoses will not be exclusive.
   * MRI findings must be normal or unremarkable for the age of the patient. Examples of abnormal (exclusory) findings are occult lacunar infarct, arteriovenous malformation) Examples of non-exclusory findings include mild atrophy, mild to moderate periventricular white matter changes. Other MRI findings will be evaluated in consultation with coinvestigator neuroradiologists and clinical judgment will be used to determine if the subject can continue in the study.

MCI Exclusion Criteria (patients):

* Other neuropsychiatric diagnoses (e.g., stroke, head trauma, any psychotic disorder, Parkinson's) other than MCI.
* Major medical illness (e.g., diabetes, severe or uncontrolled hypertension), especially potential secondary causes of cognitive decline (e.g., hypothyroidism).
* Disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image (example: coronary artery disease, hypercholesterolemia, on 5 medications, HTN 2 yrs controlled with meds, random glucose of 125, but no Dx of DM, Hx of ?TIA).
* Current substance or alcohol dependence or history of same, and no alcohol or substance abuse within the last eight weeks.

Mild Alzheimer's Disease (AD) Inclusion criteria (patients):

1. You must have a Mini Mental State Examination score of greater than 20.
2. You must have one or more of these signs and symptoms of mild AD:

Cognitive impairment manifested as memory problems, problems with language, difficulty carrying out motor activities, difficulty naming things, and/or problems planning or organizing, all of which impair function and are worsening over time.

* You must have at least 10 years of education, or a GED, or its equivalent.
* We will be drawing blood to determine your ApoE genotype. ApoE4 is a risk factor for Alzheimer's disease. We will share these results with you, if you desire to know the results. ApoE4 is only a risk factor. That means it is possible to get Alzheimer's without being ApoE4 positive, and it is possible to be ApoE4 positive and not get Alzheimer's. If you are positive for the ApoE4 genetic marker, you can be included. If you do NOT have the ApoE4 genetic marker, then you must have all other criteria.
* Age: 55-85.
* Normal or clinically unimportant physical exam, beyond those consistent with a diagnosis of mild AD.
* Able to give informed consent, or assent and informed consent from a legal representative. You will be assessed for capacity and assent/consent obtained as appropriate based on the Consensus Recommendations for Research Consent for Cognitively Impaired Adults (2004, Alzheimer's Disease Association Disorder, 18 (3):171-175).
* If you take medications that have an effect on the brain, they will be closely monitored. You will be PET-scanned only after a 24-hour washout of this medication(s), but this medication(s) will be restarted immediately after the scan.

Mild Alzheimer's Disease (AD) Exclusion Criteria:

* Any problems related to the brain or mental disorders (e.g., stroke, head trauma, any psychotic disorder, Parkinson's) other than mild AD. Some mood disorders will be acceptable because depression is often a precursor to mild AD.
* You will get an MRI of your brain taken on the second visit, and a radiologist will read it. If there are any abnormal findings, you will be told, and these findings will be forwarded to your medical doctor. These findings may or may not result in your exclusion from the study.
* Any major medical illness (e.g., diabetes, severe or uncontrolled hypertension), especially potential secondary causes of cognitive decline (e.g., hypothyroidism).
* Any disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image.
* Current diagnosis of substance or alcohol dependence or a history of same, and no alcohol or substance abuse within the last eight weeks.

MCI Inclusion criteria (controls)

* Normal cognitive screening exam.
* Age: 55-85.
* At least 10 years of education or GED, or equivalent.
* Socioeconomic status, age, and sex matched. Able to give informed consent, or assent and informed consent from a legal representative.
* Centrally acting medications will be closely tracked, patients on any such medications will be PET-scanned only after a 24-hour washout, with meds restarted immediately after the scan.

MCI Exclusion criteria (controls)

* First-degree relative with dementia or clinically relevant memory problems.
* Neuropsychiatric diagnoses (e.g., stroke, head trauma, depression, any psychoses).
* Major medical illness (e.g., diabetes, severe /uncontrolled hypertension, hypothyroidism).
* Current substance or alcohol dependence or history of same, and no alcohol or substance abuse within the last eight weeks.
* MRI findings must be normal or unremarkable for the age of the patient. Examples of abnormal (exclusory) findings are occult lacunar infarct, arteriovenous malformation) Examples of non-exclusory findings include mild atrophy, mild to moderate periventricular white matter changes. Other MRI findings will be evaluated in consultation with coinvestigator neuroradiologists and clinical judgment will be used to determine if the subject can continue in the study.

  * Disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image (example: coronary artery disease, hypercholesterolemia, on 5 medications, HTN 2 yrs controlled with meds, random glucose of 125, but no Dx of DM, Hx of ?TIA).

Dropout criteria (all):

Subjects that begin the study and are not able to finish the study will be tracked. Ongoing criteria for termination from the study will include:

* Adverse events intolerable to the patient that prevent continued involvement in the study.
* New onset medical disorder of such significance as to prohibit further involvement.
* Initiation or recurrence of alcohol or substance abuse/dependence.
* Subject withdraws consent for any reason.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must have a diagnosis of MCI or mild AD.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2003-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Determine if the Cognitive Decline Index will discriminate subtle lesions earlier than the standard analysis of the Nuclear Medicine physician. | within the next 3 years

SECONDARY OUTCOMES:
Determine if sensitivity, specificity, receiver-operator characteristics, and predictive value of our method are appropriate for translation into a clinically useful tool. | within the next three years

CONTACTS AND LOCATIONS:
Overall Officials: James Patterson, MD PhD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, Shreveport, Louisiana, United States